CLINICAL TRIAL: NCT04684888
Title: Comparison of Corneal Flap Thickness Using Visumax Femto-Lasik With SubBowman Keratomileusis (SBK) Microkeratome
Brief Title: Femto-flap Versus SBK Flap,Predictability and Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzan A Rattan (Other)
Responsible Party: Sponsor-Investigator, Suzan A Rattan, Assistant professor ophthalmologist, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10 Al-KindyCM
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Refractive Errors; Refractive Surgery
Keywords: Visumax; femtolasik; Sub Bowman keratomileusis(SBK); LASIK
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visumax Femto-flap (Active Comparator): Fifty eyes of fifty patients with age range 20-38 years, with myopic astigmatism refractive errors, ranged from -2 to- 6 DS and from -1 to -3.00DC, with stable refraction for at least one year before the surgery, normal corneal topography, anterior and posterior segments examinations. Refractive surgery was planned for both eyes and they chose the Visumax Femto-LASIK after a complete explanation of all the possible complications, costs, and differences. The right eye of each patient was taken for analysis, LASIK flap thickness was measured six months after the procedures using the anterior segment OCT, at seven points (one central and 3 points at each side of the horizontal meridian). The three nasal points were located (1mm, 2mm, 3mm respectively) from the center, and the remaining three temporal points located again ( 1mm, 2mm, 3mm) from the center.
  Interventions: Procedure: Visumax Femto-flap
- Sub Bowman's keratomileusis (SBK )-Flap group (Active Comparator): Fifty eyes of fifty patients with age range 20-38 years, with myopic astigmatism refractive errors, ranged from -2 to- 6 DS and from -1 to -3.00DC, with stable refraction for at least one year before the surgery, normal corneal topography, anterior and posterior segments examinations. They chose LASIK with mechanical SBK microkeratome surgical approach to be their refractive surgery for both eyes after all the possible complications, costs and differences had been explained clearly. The right eye of each patient was taken for analysis, LASIK flap thickness was measured six months after the procedures using the anterior segment OCT, at seven points (one central and 3 points at each side of the horizontal meridian). The three nasal points were located (1mm, 2mm, 3mm respectively) from the center, and the remaining three temporal points located again ( 1mm, 2mm, 3mm) from the center.
  Interventions: Procedure: Sub Bowman's keratomileusis (SBK)-flap

INTERVENTIONS:
Procedure: Visumax Femto-flap — Under topical anesthesia [Tetracaine eye drop 0.5%]. A-90 µm thick flap was done by using Visumax femtosecond laser. The flap hinge was set to be nasally placed. A nasal-hinge flap with 90 µm thickness, 8.8 mm flap diameter, and 90º side cut angles were created with 500 kHz Visumax FSL, 160 nJ energy [Carl Zeiss, Meditec, Germany]. The sphero- cylindrical refractive corrections with optical zone 6.5 mm and ablation zone 8.0 mm were done by excimer laser operating system [Carl Zeiss, Meditec, MEL 90, Germany]. Automatic iris registration and pupil-tracking system were activated before photoablation. The patient's eyes were examined postoperatively on a slit-lamp biomicroscope and all treatments that were given for home use have been explained in terms of frequency of instillation, possible side effects, and benefits before discharging them on the same day.
  Follow up visits were scheduled clearly on printed patients' discharging cards.
  Arms: Visumax Femto-flap
Procedure: Sub Bowman's keratomileusis (SBK)-flap — Under topical anesthesia [Tetracaine eye drop 0.5%] .A-90µm flaps done using Maria one use plus SBK mechanical microkeratome with a nasal located hinge. The sphero- cylindrical refractive corrections with optical zone 6.5 mm and ablation zone 8.0 mm were done by excimer laser operating system [Carl Zeiss, Meditec, MEL 90, Germany]. Automatic iris registration and pupil-tracking system were activated before photoablation. The patient's eyes were examined postoperatively on a slit-lamp biomicroscope and all treatments that were given for home use have been explained in terms of the frequency of instillation, possible side effects, and benefits before discharging them on the same day.
  Follow up visits were scheduled clearly on printed patients' discharging cards
  .
  Arms: Sub Bowman's keratomileusis (SBK )-Flap group

SUMMARY:
Laser Insitu keratomileusis (LASIK) has become the most popular procedure for refractive error correction. Lasik flap creation is the first and critical step during LASIK surgery because of its consensual effect on a residual stromal bed, corneal biomechanics, and hence the future risk of ectasia⁴.In the current study, we compared the Visumax FSL flap thickness predictability, accuracy, and variability with the flap created by single-use Moria SBK microkeratome.

DETAILED DESCRIPTION:
Flap creation techniques have evolved from the old manual procedure of mechanical microkeratome to the automated one with the use of microkeratome and more recently to Femto-laser procedure using a variety of machines.

Authors have reported that the primary vision nearly the same despite the different methods of flap creation in the first 6 months post LASER vision correction. Others have reported that a thinner flap is associated with better primary vision and refractive outcomes. SBK (Sub Bowman Keratomileusis), is a procedure in which the Lasik flap is thinner, and has the advantage of leaving a sufficient stromal bed for safer excimer Laser ablation.

There are five types of femtosecond Laser that were already approved currently for Lasik flap creation.

The Zeiss (Visumax FSL ) which has been used in the current study uses 1043 nm, a repetition rate of 500 kHz, and 220-580 femtoseconds pulse duration. Each laser pulse produces micro-photo disruption in the tissue, contiguous few microns sized photo disruptions will create a continuous cut in the corneal tissue at precise preset position and depth.

In the current study, the Visumax flap thickness predictability, accuracy, and variability were compared with the flap created by a single-use Moria SBK microkeratome.

ELIGIBILITY:
Inclusion Criteria:

* Having refractive errors range from -2 to- 6 DS and from -1 to -3.00DC.
* They have stable refraction for at least one year prior to surgery.
* Normal topography by Placido-Scheimpflug (Sirius, Costruzione Strumenti Oftalmici, Florence, Italia) and normal corneal epithelial map by Anterior segment-OCT system (Optovue Inc, Fremont, California, USA)

Exclusion Criteria:

1. Patient with suspicious topography and or corneal epithelial map.
2. Patient with corneal pachymetry below 500µm.
3. Patients who have a history of previous ocular surgery or trauma.
4. Patient with a current or previous history of herpes simplex or herpes zoster.
5. Patient with severe dry eye, diabetes, thyrotoxicosis, and connective tissue diseases.
6. Patient with Combined ocular diseases like retinal dystrophy or glaucoma.
7. Patient with a history of contact lenses use was meant to stop the use of soft contact lenses for at least 2 weeks or hard type for at least 4 weeks before topography and other investigations were done.
8. Patient who refrains from the required follow-up visits; have been excluded from the study.

   -

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Right eye corneal flap thickness was measured by optical coherence tomography(OCT). | 6-months postoperatively
  The lasik flap thickness in the right eye in both groups were measured six months after the procedures using non touch method by anterior segment OCT without instillation of topical anaesthesia, at seven points in each eye (one central and 3 points at each sides of horizontal meridian).The three nasal points were located (1mm, 2mm, 3mm respectively) from the center and remaining three temporal points located again ( 1mm, 2mm, 3mm) from the center. Data from both groups were comparing to evaluate predictability and variability of the flap thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Rattan, lecturer, Study Director — Al-Kindy College of Medicine
Locations (1):
- Eye Speciality private hospital, Baghdad, Iraq

REFERENCES:
- [Derived] Rattan SA, Rashid RF, Mutashar MK, Nasser YAR, Anwar DS. Comparison of corneal flap thickness predictability and architecture between femtosecond laser and sub-Bowman keratomileusis microkeratome in laser in situ keratomileusis. Int Ophthalmol. 2023 May;43(5):1553-1558. doi: 10.1007/s10792-022-02551-8. Epub 2022 Oct 29. PMID 36307607